CLINICAL TRIAL: NCT01732185
Title: Genetic and Molecular Abnormalities in Congenital Cystic Adenomatoid Malformations
Acronym: MAKP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P100510; 2012-A00538-35 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Congenital Cystic Adenomatoid Malformation (CCAM)
Keywords: Congenital lung malformation; Congenital Cystic Adenomatoid Malformation; Cystic lung disease
MeSH Terms: conditions — Cystic Adenomatoid Malformation of Lung, Congenital; Cystic Disease Of Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient (Other): congenital cystic adenomatoid malformations
  Interventions: Genetic: Patient

INTERVENTIONS:
Genetic: Patient — Blood and histological samples will be done at day of the inclusion.

SUMMARY:
The aim of this study is to identify genetic abnormalities and molecular pathways associated with the occurrence of CCAM.

DETAILED DESCRIPTION:
Congenital lung malformations are rare diseases, characterized by the coexistence in the same individual of normal lung and localized lung malformation. Among these malformations, congenital cystic adenomatoid malformations (CCAM) represent the most important group, with an estimated incidence between 1/11 000 and 1/35 000 births. The precise mechanisms leading to these lung malformations remain poorly understood. This project aims to identify key genetic and/or molecular mechanisms associated with the occurrence of CCAM. CCAMs are collected during postnatal surgical resection. Parental agreement is required. A standardised histologic description of malformations is performed for each sample. Normal lung tissue at the periphery of the malformation is considered as control. Malformations will be analyzed in a systematic way by proteome and transcriptome, after laser microdissection. Somatic genetic abnormalities will also systematically be sought.

ELIGIBILITY:
Inclusion Criteria:

* Children < 8 years
* Thoracic surgery for congenital lung malformation
* Parental written consent

Exclusion Criteria:

* Children > 8 years
* Previous infection of the malformation
* Parental rebutal

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2012-10-11 (Actual); Primary Completion 2015-10-11 (Actual); Study Completion 2015-10-11 (Actual)

PRIMARY OUTCOMES:
mRNA expression | at Day 0
  Transcriptomic analysis

SECONDARY OUTCOMES:
Protein expression | at Day 0
  Proteomic expression
Somatic genetic abnormalities | at Day 0
  CGH array

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Delacourt, MD, PhD, Principal Investigator — Necker-Enfants Malades Hospital
Locations (1):
- Necker-Enfants Malades Hospital, Paris, France

REFERENCES:
- [Background] Lezmi G, Vibhushan S, Bevilaqua C, Crapart N, Cagnard N, Khen-Dunlop N, Boyle-Freyssaut C, Hadchouel A, Delacourt C. Congenital cystic adenomatoid malformations of the lung: an epithelial transcriptomic approach. Respir Res. 2020 Feb 4;21(1):43. doi: 10.1186/s12931-020-1306-5. PMID 32019538
- [Background] Kotecha S, Barbato A, Bush A, Claus F, Davenport M, Delacourt C, Deprest J, Eber E, Frenckner B, Greenough A, Nicholson AG, Anton-Pacheco JL, Midulla F. Antenatal and postnatal management of congenital cystic adenomatoid malformation. Paediatr Respir Rev. 2012 Sep;13(3):162-70; quiz 170-1. doi: 10.1016/j.prrv.2012.01.002. Epub 2012 Apr 25. PMID 22726873